CLINICAL TRIAL: NCT03961893
Title: Panoramic Screening by Complete Colonoscopy in the Management of Colorectal Adenomas
Acronym: G-EYE-ADR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-EYE-ADR-IPC 2016-023; 2018-A03292-53 (Other: ANSM)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Adenoma
Keywords: colonoscopy; g-eye; adenomas
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Intervention Model Description: Prospective, single-phase, two-stage, randomized phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm A: Standard colonoscopy then colonoscopy with G-EYE (Experimental): Arm A: Standard colonoscopy then colonoscopy with G-EYE
  Interventions: Device: standard colonoscope first and G-EYE
- Arm B: G-EYE colonoscopy then standard colonoscopy (Experimental): Arm B: G-EYE colonoscopy then standard colonoscopy
  Interventions: Device: G-EYE first and standard colonoscope

INTERVENTIONS:
Device: G-EYE first and standard colonoscope — Patients undergo two successive colonoscopies, first balloon-assisted colonoscopy (G-EYE device) and then standard colonoscopy
  Arms: Arm B: G-EYE colonoscopy then standard colonoscopy
Device: standard colonoscope first and G-EYE — Patients undergo two successive colonoscopies, first standard colonoscopy and then balloon-assisted colonoscopy (G-EYE device)
  Arms: Arm A: Standard colonoscopy then colonoscopy with G-EYE

SUMMARY:
Colonoscopy is the gold standard for colorectal cancer prevention by allowing the resection of superficial colorectal adenomas or adenocarcinomas. This protection, more effective in the left colon than in the right colon, is imperfect and there are some adenomas and cancers omitted during colonoscopy. The G-EYE colonoscope equipped with an integrated distal balloon would better unfold the haustrations and stabilize the endoscope. Thus, the detection rate of adenomas would be improved by this better vision. The main objective of this study is to confirm that the use of the G-EYE colonoscope allows better detection of adenomatous polyps, decrease the rate of omitted adenomes and then is more effective.

ELIGIBILITY:
Inclusion Criteria:

1. Indication of complete colonoscopy for classic indications (bleeding, abdominal pain, transit disorders) or for family and personal antecedents of adenomas or colorectal cancers with the need for endoscopic control,
2. FIT + test (current blood test for stool used for mass screening in France), PET-CT fixation,
3. Consent of participation signed,
4. Affiliation to a social security scheme, or beneficiary of such a scheme.

Exclusion Criteria:

1. Non-optimal preparation (boston score <7 or segment <2),
2. Adenomatous polyposis, familial or assimilated (juvenile, etc.),
3. Pregnant or likely to be pregnant (without effective contraception) or breastfeeding,
4. Patient in emergency or deprived of liberty or placed under the authority of a tutor,
5. Patient considered geographically socially or psychologically unable to comply with the study procedure and the medical follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Rate of missed adenomas during standard colonoscopy and balloon-assisted colonoscopy (G-EYE device) | Colonoscopy time
  Rate between the number of adenomas detected by the second examination and the number of adenomas detected by the two inspections

SECONDARY OUTCOMES:
Rate of missed advanced adenomas during standard colonoscopy and balloon-assisted colonoscopy (G-EYE device) | Colonoscopy time
  Rate between the number of advanced adenomas detected by the second examination and the number of advanced adenomas detected by the two inspections
Adenoma detected rate during standard colonoscopy and balloon-assisted colonoscopy (G-EYE device) in male and female | Colonoscopy time
  Rate between the number of detected adenomas with each endoscope and the number of colonoscopies performed in male and female
Rate of complications | Colonoscopy time and 1 month after
  Global and for each arm
Rate of missed adenomas during standard colonoscopy and balloon-assisted colonoscopy (G-EYE device) in positive fetal immunochemical test (FIT+) subgroup | Colonoscopy time
  Rate between the number of adenomas detected by the second examination and the number of adenomas detected by the two inspections in FIT+ subgroup
Adenoma detected rate during standard colonoscopy and balloon-assisted colonoscopy (G-EYE device) in FIT+ subgroup | Colonoscopy time
  Rate between the number of detected adenomas with each endoscope and the number of colonoscopies performed in FIT+ subgroup
G-EYE assistance for endoscope stabilization | Colonoscopy time
  Yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe RATONE, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No